CLINICAL TRIAL: NCT06532669
Title: Explore a New Paradigm of Active Health Management for Children Based on Health Index
Brief Title: Active Health Management for Children
Status: Not yet recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-24-004
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-05

CONDITIONS: Child Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Fetal period: from the formation of the fertilized egg until before birth, approximately 40 weeks
- Neonatal period: from the beginning of umbilical cord ligation after birth to 28 days
- Infancy period: after neonatal to 1 year of age.
- Early childhood: from 1 year old to before 3 years old.
- Pre-school age: from three years old to six years old before entering primary school
- School age: from the age of 6 to the age of 12
- Puberty: from the age of 12 to the age of 18

SUMMARY:
The purpose of this study was to develop a children's active health index based on the three main factors-the environment, lifestyle, and the physiological and behavioral traits of children of various ages. To acquire dynamic data, a prospective cohort research was carried out. Construct a dynamic digital health portrait to detect and warn children's health problems early, intervene in a timely manner, and explore a new paradigm of children's active health management.

DETAILED DESCRIPTION:
Under the guidance of the World Health Organization's (WHO) Global Strategy for Women's, Children's, and Adolescents' Health (2016-2030) and China's Child Development Programme (2021-2030), as well as the comprehension that the primary focus of medical care in the future will gradually shift from disease diagnosis and treatment to disease prevention and health management, this study will develop a children's active health index based on the three main factors-the environment, lifestyle, and the physiological and behavioral traits of children of various ages-and conduct a prospective child cohort study. Gather multi-dimensional children cohort data from many sources (medical facilities, schools, families, and communities) that covers physiological indicators, behavioral habits, dietary record, and so on. The meta-model of children's active health is built using ordinary differential equations in conjunction with digital intelligence technology, which enables real-time and all-around data collection, establishes dynamic digital health portraits for children, and dynamically monitors the health status of children as it varies over time and in response to environmental changes. The ultimate goal of this approach is to identify and warn children's health problems early on, implement timely intervention, and ultimately investigate a new paradigm of children's active health management.

ELIGIBILITY:
Inclusion Criteria:

* Age≤ 18 years old, regardless of gender.
* Subject and/or guardian agrees to participate in this trial and signs the informed consent form.

Exclusion Criteria:

* The investigator judged that the subject had poor compliance and was unable to complete the study as required.
* Inability to understand the investigator's presentation or description of this trial.
* Other conditions judged by the investigator to be unsuitable for participating in the trial, such as: acute trauma, critical condition, restlessness of the subject, etc.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The target study participants were children aged 0-18 years.
Sampling Method: Non-Probability Sample
Enrollment: 1435 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Child Health Index | 0-6 years
  Child Health Index serves as a comprehensive metric to evaluate and measure how children actively maintain, promote, and enhance their own health status through positive lifestyles and healthy behaviors, with the goal of preventing the onset of diseases and delaying their progression. This index encompasses multiple aspects, such as children's dietary habits, exercise routines, sleep quality, and mental health status.

SECONDARY OUTCOMES:
Subitem Child Health Index | 0-6 years
  Child Health Index is a comprehensive index comprised of multiple subitem child health index, designed to thoroughly capture children's performance across diverse health dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Sun, MD, Principal Investigator — Xinhua Hospital, Shanghai J iao Tong University School of Medicine